CLINICAL TRIAL: NCT04740814
Title: A Multi-Center, Open-Label Study to Evaluate the Pharmacokinetics of Certolizumab Pegol in Adults With Active Rheumatoid Arthritis Using an Electrochemiluminescent Immuno-Assay
Brief Title: A Study to Assess the Pharmacokinetics of Certolizumab Pegol in Adults With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RA0138
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Results first posted 2023-11-13 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Phase 1; Cimzia; Certolizumab pegol; Electrochemiluminescent immune-assay
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Certolizumab Pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Certolizumab pegol (Experimental): Subjects in this arm will receive doses of certolizumab pegol for the treatment of Rheumatoid Arthritis, in accordance with the US label.
  Interventions: Drug: Certolizumab pegol

INTERVENTIONS:
Drug: Certolizumab pegol — * Pharmaceutical form: Solution for injection
  * Route of administration: Subcutaneous Subjects will receive certolizumab pegol in a pre-specified sequence during the study.

SUMMARY:
The purpose of the study is to evaluate the pharmacokinetics and safety of certolizumab pegol in adults with active rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 69 years of age inclusive, at the time of signing the informed consent
* Participant must have a diagnosis of moderately-to-severely active rheumatoid arthritis (RA)
* Participant must have had an inadequate response to, or intolerance to, at least 1 disease modifying antirheumatic drug (DMARD) (nonbiologic or biologic)
* Participant has a negative interferon-gamma release assay (IGRA) at Screening
* Participant has a body mass index within the range 18.0 kg/m2 to 35.0 kg/m2 (inclusive)
* Male or female
* A female participant is eligible to participate if:

  i) she is not pregnant, ii) not breastfeeding, iii) at least one of the following conditions applies:
  1. Not a woman of childbearing potential (WOCBP) OR
  2. A WOCBP who agrees to follow the contraceptive guidance during the Treatment Period and until the Safety Follow-up (SFU) Visit

     Exclusion Criteria:
* Participant has a known hypersensitivity to any components of the study medication(including polyethylene glycol) or comparative drugs (and/or an investigational device) as stated in this protocol
* Participant has clinically significant electrocardiogram (ECG) abnormalities at Screening
* Participant has previously been exposed to certolizumab pegol (CZP)
* Participant has failed treatment with ≥1 tumor necrosis factor (TNF) α inhibitor or was a primary failure for any TNFα antagonist. A primary failure is defined as no clinical disease improvement within the first 12 weeks of treatment (study participants who demonstrated clinical response within 12 weeks of treatment and subsequently lost response after 12 weeks of treatment are eligible)
* Participant has received a live vaccination within 6 weeks prior to Screening or intends to have a live vaccination during the course of the study or within 3 months following CZP treatment in the study
* Participant has received any investigational drug or experimental procedure within 90 days prior to the first dose of IMPinvestigational medicinal product (IMP)
* Participant has a laboratory abnormality at Screening, including any of the following:

  1. >3.0x upper limit of normal (ULN) of any of the following: alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP); or >ULN total bilirubin (>1.5x ULN total bilirubin if the participant has a documented pre-study diagnosis of Gilbert's syndrome)
  2. white blood cell count <3.00x103/μL
  3. absolute neutrophil count (ANC) <1.5x103/μL
  4. lymphocyte count <500 cells/μL
  5. hemoglobin <8.5 g/dL
  6. Any other laboratory abnormality, which, in the opinion of the Investigator, will prevent the study participant from completing the study or will interfere with the interpretation of the study results

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2022-01-24 (Actual); Study Completion 2022-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (14):
- United States (14):
  - Ra0138 1009, Phoenix, Arizona
  - Ra0138 1002, Covina, California
  - Ra0138 1008, Upland, California
  - Ra0138 1015, Palm Harbor, Florida
  - Ra0138 1004, Plantation, Florida
  - Ra0138 1001, Lexington, Kentucky
  - Ra0138 1014, Rockville, Maryland
  - Ra0138 1005, Albuquerque, New Mexico
  - Ra0138 10025, Duncansville, Pennsylvania
  - Ra0138 1003, Duncansville, Pennsylvania
  - Ra0138 1016, Memphis, Tennessee
  - Ra0138 1007, Austin, Texas
  - Ra0138 1010, Dallas, Texas
  - Ra0138 1011, Tomball, Texas

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size in this trial, Individual Patient Data cannot be adequately anonymized and there is a reasonable likelihood that individual participants could be re-identified. For this reason, data from this trial cannot be shared.

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in February 2021 and concluded in June 2022.
Pre-assignment Details: The Participant Flow refers to the Safety Set.
Groups:
- Certolizumab Pegol (All Participants): Participants received subcutaneous (sc) injections of certolizumab pegol (CZP) 400 milligram (mg) as loading dose at Weeks 0, 2, and 4, followed by CZP 200 mg as maintenance dose, every 2 Weeks (Q2W), up to Week 24 of the Treatment Period.
Period: Overall Study
Arm/Group | Certolizumab Pegol (All Participants)
Started | 33
Completed | 23
Not Completed | 10
Not completed — Adverse Event | 3
Not completed — Protocol Violation | 2
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Set (SS) which consisted of all study participants enrolled who received greater than or equal to (≥) 1 injection of study medication.
Arm/Group | Certolizumab Pegol (All Participants)
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 7
  White | 25
  Missing | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 24

OUTCOME MEASURES:

1. Primary Outcome: Minimum Observed Plasma Concentration (Cmin) Post 10 Weeks of Certolizumab Pegol Dosing
Description: Cmin is the Minimum observed plasma drug concentration during a dosage interval.
Time Frame: Plasma samples were collected at Pre dose on Day 70 (Week 10), 72, 75, 77 and 80 post-Week 10 study Investigational Medicinal Product (IMP) administration, and Pre dose on Day 84 (Week 12)
Population: The Pharmacokinetic Set (PKS) included the study participants who had provided plasma samples with measurable concentrations (with recorded sampling time) on at least 1 visit, and who had no important protocol deviations affecting the PK parameters. Here, Number of participants analyzed included those participants who were evaluable for the assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (ug/mL)
Arm/Group | Certolizumab Pegol (All Participants)
Number analyzed (Participants) | 25
micrograms per milliliter (ug/mL) | 24.93 (44.9)

2. Primary Outcome: Area Under the Concentration-time Curve Over One Dosing Interval (AUC0-tau) of Certolizumab Pegol
Description: AUCtau is the area Under the plasma concentration-time curve from time zero to tau for the dosing interval following administration at Week 10.
Time Frame: Plasma samples were collected at Pre dose on Day 70 (Week 10), 72, 75, 77 and 80 post-Week 10 study IMP administration, and Pre dose on Day 84 (Week 12)
Population: The PKS included the study participants who had provided plasma samples with measurable concentrations (with recorded sampling time) on at least 1 visit, and who had no important protocol deviations affecting the PK parameters. Here, Number of participants analyzed included those participants who were evaluable for the assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*ug/mL
Arm/Group | Certolizumab Pegol (All Participants)
Number analyzed (Participants) | 24
hours*ug/mL | 11890 (39.6)

3. Secondary Outcome: Plasma Concentration of Certolizumab Pegol (CZP) During the Study
Description: Plasma samples were taken at Predose and during the study at different pre and post dose time points for all participants.
Time Frame: Predose (Day 0), Day 7, 14, 42, 70, 72, 75, 77, 80, 84, 126, and 168
Population: The PKS included the study participants who had provided plasma samples with measurable concentrations (with recorded sampling time) on at least 1 visit, and who had no important protocol deviations affecting the PK parameters. Here, Number of participants analyzed included those participants who were evaluable for the assessment and 'n' (Number analyzed) signifies participants who were evaluable at specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Certolizumab Pegol (All Participants)
Number analyzed (Participants) | 28
ug/mL
  Predose (Day 0) | NA (NA) — As pre-specified in the Statistical Analysis Plan, values Below Limit of Quantification (BLQ) were replaced by value of Lower Limit of Quantification (LLOQ) divided by 2 (=0.016 ug/mL) in calculations of Means and Coefficient of Variations (CVs). Means and CVs were only calculated if at least 2/3 of the concentrations were quantified at the respective timepoint and if n is greater than equal to 4.
  Day 7: number analyzed (Participants) | 27
  Day 7 | 38.7959 (31.2)
  Day 14: number analyzed (Participants) | 27
  Day 14 | 28.7381 (25.1)
  Day 42: number analyzed (Participants) | 26
  Day 42 | 49.7912 (42.6)
  Day 70: number analyzed (Participants) | 25
  Day 70 | 29.6138 (53.6)
  Day 72: number analyzed (Participants) | 25
  Day 72 | 35.8456 (53.0)
  Day 75: number analyzed (Participants) | 25
  Day 75 | 38.8787 (42.2)
  Day 77: number analyzed (Participants) | 23
  Day 77 | 37.4564 (38.1)
  Day 80: number analyzed (Participants) | 23
  Day 80 | 33.9728 (39.1)
  Day 84: number analyzed (Participants) | 24
  Day 84 | 27.9509 (45.9)
  Day 126: number analyzed (Participants) | 24
  Day 126 | 21.2735 (129.1)
  Day 168: number analyzed (Participants) | 22
  Day 168 | 22.9050 (46.6)

4. Secondary Outcome: Percentage of Participants With Treatment-emergent Serious Adverse Event (SAEs)
Description: A treatment-emergent adverse event (TEAE) was defined as events that have a start date on or following the first administration of study treatment in this study through the final administration of study treatment+70 days through Safety Follow-up (SFU) visit. A Serious Adverse Event (SAE) is any untoward medical occurrence that at any dose: Results in death, Is life-threatening, Requires in patient hospitalization or prolongation of existing hospitalization, Results in persistent disability/incapacity, Is a congenital anomaly or birth defect, Other important medical events which based on medical or scientific judgement may jeopardize the patients, or may require medical or surgical intervention to prevent any of the above.
Time Frame: From Baseline to the Safety Follow-up Visit (up to Week 34)
Population: The SS included all study participants enrolled who received ≥1 injection of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Certolizumab Pegol (All Participants)
Number analyzed (Participants) | 33
percentage of participants | 6.1

5. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Event (TEAEs) Leading to Withdrawal
Description: An Adverse event (AE) was any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study medication, whether or not considered related to the study medication. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study medication. A TEAE was defined as events that have a start date on or following the first administration of study treatment in this study through the final administration of study treatment+70 days through Safety Follow-up (SFU) visit.
Time Frame: From Baseline to the Safety Follow-up Visit (up to Week 34)
Population: The SS included all study participants enrolled who received ≥1 injection of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Certolizumab Pegol (All Participants)
Number analyzed (Participants) | 33
percentage of participants | 9.1

ADVERSE EVENTS:
Time Frame: From Screening to the Safety Follow-up Visit (up to 38 Weeks)
Description: An AE was any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study medication, whether or not considered related to the study medication. The SS included all study participants enrolled who received ≥1 injection of study medication. All AEs from Screening until the End of study are reported here.
Arm/Group | Certolizumab Pegol (All Participants)
All-Cause Mortality (participants affected / at risk) | 1/33
Serious Adverse Events (participants affected / at risk) | 2/33
Other Adverse Events (participants affected / at risk) | 9/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Certolizumab Pegol (All Participants) (N=33)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Certolizumab Pegol (All Participants) (N=33)
Nausea (Gastrointestinal disorders) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 3 (3)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-03-18): https://cdn.clinicaltrials.gov/large-docs/14/NCT04740814/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-30): https://cdn.clinicaltrials.gov/large-docs/14/NCT04740814/SAP_001.pdf